CLINICAL TRIAL: NCT02331914
Title: Gastrointestinal Stromal Tumors: Assessment of Mutations in Tumors and in Circulating Tumor DNA and Measurement of TKI Plasma Exposure to Optimize Treatment
Brief Title: GIST: Assessment of Tumor Mutations and TKI Plasma Exposure
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: 19082014
Record Dates: First submitted 2014-12-29; First posted 2015-01-06 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Gastro-intestinal Stromal Tumor
Keywords: GIST; Bio-databank

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor biopsy after disease progression
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gastro-intestinal stromal tumors: A bio-databank consisting of TKI drug level and serum for analysis of mutations in circulating tumor DNA will be set up. This bio-databank will be used to study whether changes in the amount of the primary KIT mutation is an early predictor of treatment response and/of failure. Moreover, secondary TKI resistant mutations in circulating tumor DNA will be assessed.
  To be able to assess those mutations, a tumor biopsy will be performed at the time of radiologic progressive disease. Vena puncture for blood collection will be performed at routine out patient visits.
  Interventions: Procedure: Vena puncture for blood collection; Procedure: Tumor biopsy

INTERVENTIONS:
Procedure: Vena puncture for blood collection — GIST patients will be asked to provide 40ml blood that will be collected in four Na-EDTA 10ml blood collection tubes at every routine outpatient visit.
Procedure: Tumor biopsy — Tumor biopsy after disease progression

SUMMARY:
Gastrointestinal stromal tumors (GISTs) belong to the sarcoma group and are characterized by oncogenic mutations in the c-KIT, PDGFRA, BRAF and NF-1 genes that drive tumor growth. Since tyrosine kinase inhibitors (TKIs) have become available, the median survival of GIST patients increased from 9 months to over 5 years. Consequently, this rare disease has become a role model for other targeted therapies. However, response to TKIs is extremely heterogeneous: ~15% of the patients experience no benefit from imatinib, whereas ~17% of the patients enjoy stable disease for over 9 years. Treatment failure due to primary and secondary resistance is caused in part by mutations in oncogenic genes that cause change in drug sensitivity. A new technique, using circulating tumor DNA, has enabled us to assess mutations in a simple blood sample obtained from patients on treatment, and thus detect new mutations early in the course of the disease. Also, differences in pharmacokinetic drug behavior add to the observed heterogeneity, and may cause resistance due to drug underexposure and thereby proliferation of the least sensitive tumor cells. This offers the opportunity to optimize and personalize targeted treatment for individual GIST patients by timely treatment adaptation based on early detection of secondary TKIs resistance mutations. Achieving this urgently requires data on daily clinical practice, including prospective serial mutation analysis and serial drug plasma concentration measurement. At a fundamental level this will also help to unravel the driving factors behind primary and secondary TKIs resistance in this model disease.

DETAILED DESCRIPTION:
The treatment of Dutch GIST patients is centralized: almost all patients are referred to one of the five collaborating centers forming the Dutch GIST consortium, UMCG, NKI-AvL, Radboud UMC, Erasmus MC and LUMC. To further optimize treatment for all patients, these centers have implemented a standard-of-care diagnostic and treatment plan that assures collection of homogenous phenotypic and treatment data for the bio-databank. The consortium is supported by and works in close collaboration with the Dutch sarcoma and GIST patient organizations.

A prospective, longitudinal bio-databank will be set up. Data regarding multi-morbidity, drug pharmacokinetics and serial tumor genotypic data will be collected prospectively from all (new) GIST patients during TKI treatment. Our standard-of-care plan includes primary tumor mutation analysis, performed by pathology laboratories on site. At each follow up visit during treatment, blood will be collected to assess TKI plasma exposure and to perform mutation analysis on circulating tumor DNA. All patients will be followed for tumor RECIST 1.1 progression assessed by CT scans and asked to undergo a tumor biopsy at progression to detect secondary resistance mutations.

The development of a model predicting secondary imatinib resistance based on patient phenotype and tumor genotype, will be achieved by analyzing GIST patients with progressive disease on imatinib (index patients; n=30) in our bio-databank. These patients will be matched 1:1 with non-progressive patients treated for the same duration as the index patients. Regarding the index patients, next-generation gene-targeted mutation analysis will be performed on archival tumor material and on a tumor biopsy at progression to identify patient's unique secondary mutations. The mutations that will be studied are: KIT exon 9, exon 11, exon 13, exon 14, exon 17 and exon 18; PDGFRA exon 12, exon 14 and exon 18 and BRAF exon 10 en exon 15.

In-depth analysis regarding mutation analysis in circulating tumor DNA and imatinib drug concentration assessment will be performed for these 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a GIST with an indication to be treated with a TKI of whom a histological biopsy before start treatment is available.
* Informed consent is given

Exclusion Criteria:

* Patients of whom no tumor is available before start of first line TKI
* Patients that refuse a tumor biopsy in case of tumor progression
* Patients in whom it will not be possible to perform a biopsy in case of tumor progression (for example anti-coagulants that cannot be interrupted).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic gastrointestinal stromal tumors treated with tyrosine kinase inhibitors.
Sampling Method: Probability Sample
Enrollment: 740 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Secondary GIST mutations in circulating tumor DNA of patients with progressive disease on TKI treatment | 2 years
  To assess whether secondary GIST mutations can be found in circulating tumor DNA of patients with progressive disease on TKI treatment (according to RECIST 1.1 on computer tomography), whereas they are NOT present in the patients that have no progressive disease after the same time of TKI treatment

SECONDARY OUTCOMES:
Secondary mutations in circulating tumor DNA before progressive disease according RECIST | 2 years
  To establish whether these secondary mutations can be detected some time (> 3 months) before progressive disease is assessed according to RECIST 1.1 on computer tomography
Secondary mutations in circulating tumor DNA related to pharmacokinetics of TKI | 2 years
  To assess whether the occurence of secondary mutations in circulating tumor DNA is related to TKI trough levels

CONTACTS AND LOCATIONS:
Overall Officials: A. K. Reyners, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (5):
- Netherlands (5):
  - Antoni van Leeuwenhoek Hospital, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - University Medical Center St. Radboud, Nijmegen
  - Erasmus MC, Rotterdam